CLINICAL TRIAL: NCT03654105
Title: Multifactorial Intervention of Primary Prevention in High Risk Subjects: a Randomized Trial
Brief Title: Screening and Multiple Intervention on Lung Epidemics
Acronym: SMILE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: Istituto Di Ricerche Farmacologiche Mario Negri (Other)
Responsible Party: Principal Investigator, Ugo Pastorino, Head of Thoracic Surgery Division, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 2016-003036-20
Record Dates: First submitted 2018-08-14; First posted 2018-08-31 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Inflammation; Smoking Cessation; Diet Modification; Physical Activity; Lung Cancer
Keywords: Inflammation; Primary Prevention; Multiple Prevention; Lung Cancer Screening; Smoking Cessation; Diet; Physical Activity; CRP
MeSH Terms: conditions — Inflammation; Smoking Cessation; Motor Activity; Lung Neoplasms | interventions — cytisine; Aspirin; Diet Therapy; Spirometry; Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Smoking cessation and Antinflammatory (Experimental): Smoking cessation through the administration of Cytisine (in standard and prolonged administration) + reduction of inflammatory status through the administration of Acetylsalicylic acid, diet modification and physical activity increase + standard treatment for early lung cancer detection (ultra low dose CT) + spirometry with CO test + anthropometic data collection + blood test
  Interventions: Drug: Cytisine; Drug: Acetylsalicylic acid; Other: Diet Modification and Physical Activity Increase; Diagnostic Test: early lung cancer detection; Diagnostic Test: spirometry with CO test; Other: anthropometic data collection; Other: blood test
- Smoking cessation (Experimental): Smoking cessation through the administration of Cytisine (in standard and prolonged administration) + standard treatment for early lung cancer detection (ultra low dose CT) + spirometry with CO test + anthropometic data collection + blood test
  Interventions: Drug: Cytisine; Diagnostic Test: early lung cancer detection; Diagnostic Test: spirometry with CO test; Other: anthropometic data collection; Other: blood test
- Antinflammatory (Experimental): reduction of inflammatory status through the administration of Acetylsalicylic acid, diet modification and physical activity increase + standard treatment for early lung cancer detection (ultra low dose CT) + spirometry with CO test + anthropometic data collection + blood test
  Interventions: Drug: Acetylsalicylic acid; Other: Diet Modification and Physical Activity Increase; Diagnostic Test: early lung cancer detection; Diagnostic Test: spirometry with CO test; Other: anthropometic data collection; Other: blood test
- Control Group (Other): standard treatment for early lung cancer detection (ultra low dose CT) + spirometry with CO test + anthropometic data collection + blood test
  Interventions: Diagnostic Test: early lung cancer detection; Diagnostic Test: spirometry with CO test; Other: anthropometic data collection; Other: blood test

INTERVENTIONS:
Drug: Cytisine — Cytisine administration will be randomized 1:1 in standard (40 days)and prolonged treatment (84 days).
  Subjects will be educated on how to take the product and informed about possible adverse effects.
  Other Names: ev code SUB31171
  Arms: Smoking cessation; Smoking cessation and Antinflammatory
Drug: Acetylsalicylic acid — The treatment will consist of Acetylsalicylic acid at 100mg once a day
  Other Names: Cardioaspirin
  Arms: Antinflammatory; Smoking cessation and Antinflammatory
Other: Diet Modification and Physical Activity Increase — It will be proposed:
  1. an optimal diet with the aim of favoring control of weight, abdominal fat and adequate nutritional status without increasing the levels of IGF-I and inflammatory factors or glycemic peaks, with periodic verification of the results
  2. a regular and sustainable physical activity program with periodic verification of the results.
  Arms: Antinflammatory; Smoking cessation and Antinflammatory
Diagnostic Test: early lung cancer detection — standard treatment for early lung cancer detection with ultra low dose CT
Diagnostic Test: spirometry with CO test — spirometry with CO test
Other: anthropometic data collection — anthropometic data collection
Other: blood test — blood test to assess the metabolic and inflammatory profile

SUMMARY:
This prospective randomized pilot trial will evaluate a multiple intervention program of prevention in lifelong smokers aiming at reduction of chronic inflammation status through treatment with low-dose acetylsalicylic acid (ASA), smoking cessation with cytisine, targeted modification of diet and physical activity, in addition to early diagnosis with annual ultra low-dose spiral computed tomography (LDCT).

DETAILED DESCRIPTION:
The most recent population-based studies carried out in Europe and the US on hundreds of thousands of individuals have unequivocally identified three principal causes of mortality, morbidity and chronic disability: tobacco smoke, inadequate diet, and reduced physical activity. These risk factors are in large part reversible, because in heavy smokers, even after 60 years of age, cessation is associated with a clear reduction in all-cause mortality. The finding that lifestyle and eating habits are associated with the development of cancer has been confirmed in many studies: smoking, a sedentary lifestyle, excess red meat, processed foods and sugars are associated with increased risk, while an active lifestyle, non-exposure to smoke (both active and passive), consumption of whole grains, legumes and vegetables are associated with protection or a reduced incidence in at-risk subjects.

What is clear, and confirmed by many studies, is that cancer occurs more often in overweight individuals, and that cancer patients who are overweight have more difficulty treating their disease. Elevated plasma levels of C-reactive protein (CRP), even when still within normal limits, are the reflection of a chronic state of inflammation and are associated with poor prognosis in several tobacco-related diseases. CRP measurement is besides a simple test to predict the risk of heart attack and stroke as well as mortality from all causes and from cardiovascular disease. In a systematic review on adult solid tumors, elevated CRP levels were associated with higher mortality and recurrence rates, and this observation was confirmed in early-stage lung cancer by a recent meta-analysis. In patients with chronic obstructive pulmonary disease (COPD), high CRP is a strong and independent predictor of future morbidity and mortality, and an increase in CRP concurrent with a reduction of the forced expiratory volume in 1 second (FEV1) shows an even stronger effect on patient's outcome.

High levels of CRP are associated with poor prognosis in cancers of the upper aerodigestive tract, rhinopharynx, lung and urinary tract. From a dietary point of view, consumption of saturated fats has been directly associated with an increase in inflammatory status as measured by high levels of CRP, just like consumption of meat, while an inverse correlation with consumption of vegetables has been observed. For example, low levels of inflammatory factors have been found in individuals adhering to a Mediterranean diet. Another recurrent finding, at least for cancer, is the importance of daily physical activity, such as brisk walking for 30 minutes. Moreover, regular physical activity is associated with better prognosis and increased survival in patients with a cancer diagnosis.

The number of heavy smokers that will participate in early-diagnosis programs using spiral CT will undoubtedly increase in the future as a result of awareness campaigns, and the participating volunteers represent an excellent opportunity to evaluate the efficacy of targeted primary prevention programs.

The present program will combine several interventions according to the randomization arm, proposed in combination or in single treatment, including treatment with cytisine, reduction of chronic inflammation by treatment with low-dose aspirin (ASA), targeted modification of diet and physical activity, in addition to early diagnosis with annual ultra low-dose spiral computed tomography (LDCT).

At baseline each volunteer will undergo:

* questionnaires on population evaluation (e.g. socio-demographic, smoking habits, physical activity, etc)
* blood sampling for the assessment of the inflammatory and metabolic profile
* evaluation of respiratory function and measurement of carbon monoxide (CO)
* thorax ultra low-dose computed tomography (LDCT) without contrast
* anthropometric evaluation (e.g. weight, height, BMI, etc)

To reduce levels of chronic inflammation will be used:

* treatment with low-dose acetylsalicylic acid (ASA)
* dietary / nutritional intervention in order to promote an optimal diet, based on characteristic of the Mediterranean Diet, for weight maintenance, visceral fat control and an adequate nutritional status
* physical activity intervention, through the reduction of sedentary behaviour and the implementation of a moderate intensity activity of about 30 min a day

In the Smoking cessation will be used Cytisine. It is a molecule known since the early 60s for the treatment of smoking. In recent clinical trials it revealed efficacy in smoking cessation. In 2014, the NHS (National Health Service) produced a document evaluating the cost-effectiveness of drug treatment of smoking, concluding that cytisine has the most favorable profile among the drugs taken into consideration

The imaging will be performed by volumetric acquisition with a computed tomography scanner equipped with advanced technology hardware and software, including: high performance X-ray tube with low potential, high sensitivity detectors combined with dedicated reconstruction algorithms for optimisation of the signal to noise ratio within an ultra low radiation dose. The protocol for ultra-low dose computed tomography will be specifically set for lung cancer screening with semiautomated image analysis and nodule quantification, according to the international standard for image quality (Quantitative Imaging Biomarker Alliance). In particular, the ultra-low dose computed tomography protocol will be developed for the lowest radiation exposure and tested by dedicated phantom for quantitative analysis of imaging metrics.

In the control group subjects will receive an information booklet containing advice on an optimal lifestyle with particular reference to smoking, diet and physical activity according to the best international guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Age between 55 and 75 years
* High consumption of cigarettes (≥ 30 packs/year)
* Elegibility to annual LDCT screening
* Confidence in Internet use
* Absence of tumors for at least 5 years
* Signed informed consent form

Exclusion Criteria:

* Hypersensitivity to acetylsalicylic acid, salicylates or any of the excipients (excipients: cellulose powder, corn starch, coating: copolymers of methacrylic acid, sodium lauryl sulfate, polysorbate 80, talc, triethyl citrate)
* Chronic treatment with acetylsalicylic acid, or other anti-clotting or anti-coagulant drugs (for example: heparin, dicumarol)
* Treatment with methotrexate
* Existing Mastocytosis
* History of asthma induced by the administration of salicylates or substances to similar activity, particularly non-steroidal anti-inflammatory drugs
* Gastroduodenal ulcer
* Hemorrhagic diathesis
* Severe chronic pathology (eg: severe respiratory and / or renal and / or hepatic and / or cardiac insufficiency)
* Serious psychiatric problems
* Previous treatment with Cytisine
* Abuse of alcohol or other substances (even previous)

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2019-07-23 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in chronic inflammatory status | 1 year
  Reduction in the percentage of subjects with CRP>=2 mg/L

SECONDARY OUTCOMES:
Change in smoking status | 1 year
  Reduction in the percentage of smokers
Change in dietary habits | 1 year
  Dietary intakes are collected by a self reported food frequencies questionnaire and data are expressed as the average daily/weekly consumption of foods and food groups.
  Servings size is defined as "natural unit" (e.g. 1 glass of soft drinks, 1 teaspoon of sugar) or as an average serving (e.g. 80 g of pasta or rice, 30 g of dried fruits).
  The frequency of serving size is reported as continuous measure. Data will be collected as continuous measures and will be analyzed by performing statistical models to investigate a potential relationship among changes in dietary habits and anthropometric parameters (BMI, waist circumference..), socio-demographic characteristics (gender, smoking status, physical activity), biochemical parameters (CRP blood levels), drugs assumption and the risk of chronic diseases, such as lung cancer.
Change in the physical activity | 1 year
  Increase in the physical activity measured by the validate short form IPAQ questionnaire (International Physical Activity Questionnaire) The items in the short IPAQ form were structured to provide separate scores on walking, moderate-intensity and vigorous-intensity activity. Computation of the total score requires summation of the duration (in minutes) and frequency (days) of each activity.
  METs are multiples of the resting metabolic rate and a MET-minute is computed by multiplying the MET score of an activity by the minutes performed:
  * Walking MET-minutes/week = 3.3 * walking minutes * walking days
  * Moderate MET-minutes/week = 4.0 * moderate-intensity activity minutes * moderate days
  * Vigorous MET-minutes/week = 8.0 * vigorous-intensity activity minutes * vigorous-intensity days
  * Total physical activity MET-minutes/week = sum of Walking + Moderate + Vigorous MET-minutes/week scores
Change in body mass index (BMI) | 1 year
  Weight and height will be combined to report BMI in kg/m^2. Reduction in BMI
Change in waist circumference | 1 year
  Reduction in waist circumference expressed in centimeters
Change in metabolic profile | 1 year
  Enhancement in blood glucose, total cholesterol, LDL, HDL and triglycerides
Change in lung cancer incidence | 3 years
  Reduction in lung cancer incidence
Change in lung cancer specific and overall mortality | 3 years
  Reduction in lung cancer specific and overall mortality

CONTACTS AND LOCATIONS:
Overall Officials: Ugo Pastorino, MD, Principal Investigator — IRCCS IstitutoNazionale dei Tumori di Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pastorino U, Boffi R, Marchiano A, Sestini S, Munarini E, Calareso G, Boeri M, Pelosi G, Sozzi G, Silva M, Sverzellati N, Galeone C, La Vecchia C, Ghirardi A, Corrao G. Stopping Smoking Reduces Mortality in Low-Dose Computed Tomography Screening Participants. J Thorac Oncol. 2016 May;11(5):693-699. doi: 10.1016/j.jtho.2016.02.011. Epub 2016 Feb 24. PMID 26921675
- [Background] Pastorino U, Morelli D, Marchiano A, Sestini S, Suatoni P, Taverna F, Boeri M, Sozzi G, Cantarutti A, Corrao G. Inflammatory status and lung function predict mortality in lung cancer screening participants. Eur J Cancer Prev. 2018 Jul;27(4):289-295. doi: 10.1097/CEJ.0000000000000342. PMID 28333763
- [Background] Pastorino U, Morelli D, Leuzzi G, Gisabella M, Suatoni P, Taverna F, Bertocchi E, Boeri M, Sozzi G, Cantarutti A, Corrao G. Baseline and postoperative C-reactive protein levels predict mortality in operable lung cancer. Eur J Cancer. 2017 Jul;79:90-97. doi: 10.1016/j.ejca.2017.03.020. Epub 2017 May 1. PMID 28472743
- [Background] La Vecchia C, Gallus S, Garattini S. Effects of physical inactivity on non-communicable diseases. Lancet. 2012 Nov 3;380(9853):1553; author reply 1553-4. doi: 10.1016/S0140-6736(12)61872-8. No abstract available. PMID 23122239
- [Background] Bonaccio M, Cerletti C, Iacoviello L, de Gaetano G. Mediterranean diet and low-grade subclinical inflammation: the Moli-sani study. Endocr Metab Immune Disord Drug Targets. 2015;15(1):18-24. doi: 10.2174/1871530314666141020112146. PMID 25329200
- [Background] Lee Y, Kang D, Lee SA. Effect of dietary patterns on serum C-reactive protein level. Nutr Metab Cardiovasc Dis. 2014 Sep;24(9):1004-11. doi: 10.1016/j.numecd.2014.05.001. Epub 2014 May 27. PMID 24998076
- [Background] Bosetti C, Gallus S, Peto R, Negri E, Talamini R, Tavani A, Franceschi S, La Vecchia C. Tobacco smoking, smoking cessation, and cumulative risk of upper aerodigestive tract cancers. Am J Epidemiol. 2008 Feb 15;167(4):468-73. doi: 10.1093/aje/kwm318. Epub 2007 Dec 4. PMID 18056925
- [Background] Gallus S, Muttarak R, Martinez-Sanchez JM, Zuccaro P, Colombo P, La Vecchia C. Smoking prevalence and smoking attributable mortality in Italy, 2010. Prev Med. 2011 Jun;52(6):434-8. doi: 10.1016/j.ypmed.2011.03.011. Epub 2011 Mar 21. PMID 21421001
- [Background] Linseisen J, Rohrmann S, Miller AB, Bueno-de-Mesquita HB, Buchner FL, Vineis P, Agudo A, Gram IT, Janson L, Krogh V, Overvad K, Rasmuson T, Schulz M, Pischon T, Kaaks R, Nieters A, Allen NE, Key TJ, Bingham S, Khaw KT, Amiano P, Barricarte A, Martinez C, Navarro C, Quiros R, Clavel-Chapelon F, Boutron-Ruault MC, Touvier M, Peeters PH, Berglund G, Hallmans G, Lund E, Palli D, Panico S, Tumino R, Tjonneland A, Olsen A, Trichopoulou A, Trichopoulos D, Autier P, Boffetta P, Slimani N, Riboli E. Fruit and vegetable consumption and lung cancer risk: updated information from the European Prospective Investigation into Cancer and Nutrition (EPIC). Int J Cancer. 2007 Sep 1;121(5):1103-14. doi: 10.1002/ijc.22807. PMID 17487840
- [Background] Lugo A, Asciutto R, Pacifici R, Colombo P, La Vecchia C, Gallus S. Smoking in Italy 2013-2014, with a focus on the young. Tumori. 2015 Sep-Oct;101(5):529-34. doi: 10.5301/tj.5000311. Epub 2015 May 15. PMID 25983096
- [Background] Peto J. Cancer epidemiology in the last century and the next decade. Nature. 2001 May 17;411(6835):390-5. doi: 10.1038/35077256. PMID 11357148
- [Background] Lee IM, Shiroma EJ, Lobelo F, Puska P, Blair SN, Katzmarzyk PT; Lancet Physical Activity Series Working Group. Effect of physical inactivity on major non-communicable diseases worldwide: an analysis of burden of disease and life expectancy. Lancet. 2012 Jul 21;380(9838):219-29. doi: 10.1016/S0140-6736(12)61031-9. PMID 22818936
- [Background] Carter BD, Abnet CC, Feskanich D, Freedman ND, Hartge P, Lewis CE, Ockene JK, Prentice RL, Speizer FE, Thun MJ, Jacobs EJ. Smoking and mortality--beyond established causes. N Engl J Med. 2015 Feb 12;372(7):631-40. doi: 10.1056/NEJMsa1407211. PMID 25671255
- [Background] Muezzinler A, Mons U, Gellert C, Schottker B, Jansen E, Kee F, O'Doherty MG, Kuulasmaa K, Freedman ND, Abnet CC, Wolk A, Hakansson N, Orsini N, Wilsgaard T, Bueno-de-Mesquita B, van der Schouw YT, Peeters PHM, de Groot LCPGM, Peters A, Orfanos P, Linneberg A, Pisinger C, Tamosiunas A, Baceviciene M, Luksiene D, Bernotiene G, Jousilahti P, Petterson-Kymmer U, Jansson JH, Soderberg S, Eriksson S, Jankovic N, Sanchez MJ, Veronesi G, Sans S, Drygas W, Trichopoulou A, Boffetta P, Brenner H. Smoking and All-cause Mortality in Older Adults: Results From the CHANCES Consortium. Am J Prev Med. 2015 Nov;49(5):e53-e63. doi: 10.1016/j.amepre.2015.04.004. Epub 2015 Jul 15. PMID 26188685
- [Background] Thun MJ, Carter BD, Feskanich D, Freedman ND, Prentice R, Lopez AD, Hartge P, Gapstur SM. 50-year trends in smoking-related mortality in the United States. N Engl J Med. 2013 Jan 24;368(4):351-64. doi: 10.1056/NEJMsa1211127. PMID 23343064
- [Background] Doll R, Peto R, Boreham J, Sutherland I. Mortality in relation to smoking: 50 years' observations on male British doctors. BMJ. 2004 Jun 26;328(7455):1519. doi: 10.1136/bmj.38142.554479.AE. Epub 2004 Jun 22. PMID 15213107
- [Background] Peto R, Darby S, Deo H, Silcocks P, Whitley E, Doll R. Smoking, smoking cessation, and lung cancer in the UK since 1950: combination of national statistics with two case-control studies. BMJ. 2000 Aug 5;321(7257):323-9. doi: 10.1136/bmj.321.7257.323. PMID 10926586
- [Background] Gallus S, La Vecchia C, Levi F, Simonato L, Dal Maso L, Franceschi S. Leanness and squamous cell oesophageal cancer. Ann Oncol. 2001 Jul;12(7):975-9. doi: 10.1023/a:1011104809985. PMID 11521805
- [Background] Franceschi S, Dal Maso L, Levi F, Conti E, Talamini R, La Vecchia C. Leanness as early marker of cancer of the oral cavity and pharynx. Ann Oncol. 2001 Mar;12(3):331-6. doi: 10.1023/a:1011191809335. PMID 11332144
- [Background] Duan P, Hu C, Quan C, Yi X, Zhou W, Yuan M, Yu T, Kourouma A, Yang K. Body mass index and risk of lung cancer: Systematic review and dose-response meta-analysis. Sci Rep. 2015 Nov 19;5:16938. doi: 10.1038/srep16938. PMID 26582414
- [Background] Kabat GC, Kim M, Hunt JR, Chlebowski RT, Rohan TE. Body mass index and waist circumference in relation to lung cancer risk in the Women's Health Initiative. Am J Epidemiol. 2008 Jul 15;168(2):158-69. doi: 10.1093/aje/kwn109. Epub 2008 May 15. PMID 18483121
- [Background] Lam TK, Moore SC, Brinton LA, Smith L, Hollenbeck AR, Gierach GL, Freedman ND. Anthropometric measures and physical activity and the risk of lung cancer in never-smokers: a prospective cohort study. PLoS One. 2013 Aug 5;8(8):e70672. doi: 10.1371/journal.pone.0070672. Print 2013. PMID 23940620
- [Background] Etemadi A, O'Doherty MG, Freedman ND, Hollenbeck AR, Dawsey SM, Abnet CC. A prospective cohort study of body size and risk of head and neck cancers in the NIH-AARP diet and health study. Cancer Epidemiol Biomarkers Prev. 2014 Nov;23(11):2422-9. doi: 10.1158/1055-9965.EPI-14-0709-T. Epub 2014 Aug 29. PMID 25172872
- [Background] Gaudet MM, Kitahara CM, Newton CC, Bernstein L, Reynolds P, Weiderpass E, Kreimer AR, Yang G, Adami HO, Alavanja MC, Beane Freeman LE, Boeing H, Buring J, Chaturvedi A, Chen Y, D'Aloisio AA, Freedman M, Gao YT, Gaziano JM, Giles GG, Hakansson N, Huang WY, Lee IM, Linet MS, MacInnis RJ, Park Y, Prizment A, Purdue MP, Riboli E, Robien K, Sandler DP, Schairer C, Sesso HD, Ou Shu X, White E, Wolk A, Xiang YB, Zelenuich-Jacquotte A, Zheng W, Patel AV, Hartge P, Berrington de Gonzalez A, Gapstur SM. Anthropometry and head and neck cancer:a pooled analysis of cohort data. Int J Epidemiol. 2015 Apr;44(2):673-81. doi: 10.1093/ije/dyv059. Epub 2015 Jun 6. PMID 26050257
- [Background] Anandavadivelan P, Lagergren P. Cachexia in patients with oesophageal cancer. Nat Rev Clin Oncol. 2016 Mar;13(3):185-98. doi: 10.1038/nrclinonc.2015.200. Epub 2015 Nov 17. PMID 26573424
- [Background] Andersson BA, Lewin F, Lundgren J, Nilsson M, Rutqvist LE, Lofgren S, Laytragoon-Lewin N. Plasma tumor necrosis factor-alpha and C-reactive protein as biomarker for survival in head and neck squamous cell carcinoma. J Cancer Res Clin Oncol. 2014 Mar;140(3):515-9. doi: 10.1007/s00432-014-1592-8. Epub 2014 Jan 31. PMID 24481866
- [Background] Xia WX, Ye YF, Lu X, Wang L, Ke LR, Zhang HB, Roycik MD, Yang J, Shi JL, Cao KJ, Guo X, Xiang YQ. The impact of baseline serum C-reactive protein and C-reactive protein kinetics on the prognosis of metastatic nasopharyngeal carcinoma patients treated with palliative chemotherapy. PLoS One. 2013 Oct 10;8(10):e76958. doi: 10.1371/journal.pone.0076958. eCollection 2013. PMID 24130817
- [Background] Hong S, Kang YA, Cho BC, Kim DJ. Elevated serum C-reactive protein as a prognostic marker in small cell lung cancer. Yonsei Med J. 2012 Jan;53(1):111-7. doi: 10.3349/ymj.2012.53.1.111. PMID 22187240
- [Background] Dai J, Tang K, Xiao W, Yu G, Zeng J, Li W, Zhang YQ, Xu H, Chen ZQ, Ye ZQ. Prognostic significance of C-reactive protein in urological cancers: a systematic review and meta-analysis. Asian Pac J Cancer Prev. 2014;15(8):3369-75. doi: 10.7314/apjcp.2014.15.8.3369. PMID 24870724
- [Background] Santos S, Oliveira A, Lopes C. Systematic review of saturated fatty acids on inflammation and circulating levels of adipokines. Nutr Res. 2013 Sep;33(9):687-95. doi: 10.1016/j.nutres.2013.07.002. Epub 2013 Aug 6. PMID 24034567
- [Background] Trichopoulou A, Kouris-Blazos A, Wahlqvist ML, Gnardellis C, Lagiou P, Polychronopoulos E, Vassilakou T, Lipworth L, Trichopoulos D. Diet and overall survival in elderly people. BMJ. 1995 Dec 2;311(7018):1457-60. doi: 10.1136/bmj.311.7018.1457. PMID 8520331
- [Background] Montgomery AA, Peters TJ, Little P. Design, analysis and presentation of factorial randomised controlled trials. BMC Med Res Methodol. 2003 Nov 24;3:26. doi: 10.1186/1471-2288-3-26. PMID 14633287
- [Background] Pastorino U, Bellomi M, Landoni C, De Fiori E, Arnaldi P, Picchio M, Pelosi G, Boyle P, Fazio F. Early lung-cancer detection with spiral CT and positron emission tomography in heavy smokers: 2-year results. Lancet. 2003 Aug 23;362(9384):593-7. doi: 10.1016/S0140-6736(03)14188-8. PMID 12944057
- [Background] Global BMI Mortality Collaboration, Di Angelantonio E, Bhupathiraju ShN, Wormser D, Gao P, Kaptoge S, Berrington de Gonzalez A, Cairns BJ, Huxley R, Jackson ChL, Joshy G, Lewington S, Manson JE, Murphy N, Patel AV, Samet JM, Woodward M, Zheng W, Zhou M, Bansal N, Barricarte A, Carter B, Cerhan JR, Smith GD, Fang X, Franco OH, Green J, Halsey J, Hildebrand JS, Jung KJ, Korda RJ, McLerran DF, Moore SC, O'Keeffe LM, Paige E, Ramond A, Reeves GK, Rolland B, Sacerdote C, Sattar N, Sofianopoulou E, Stevens J, Thun M, Ueshima H, Yang L, Yun YD, Willeit P, Banks E, Beral V, Chen Zh, Gapstur SM, Gunter MJ, Hartge P, Jee SH, Lam TH, Peto R, Potter JD, Willett WC, Thompson SG, Danesh J, Hu FB. Body-mass index and all-cause mortality: individual-participant-data meta-analysis of 239 prospective studies in four continents. Lancet. 2016 Aug 20;388(10046):776-86. doi: 10.1016/S0140-6736(16)30175-1. Epub 2016 Jul 13. PMID 27423262
- [Background] West R, Zatonski W, Cedzynska M, Lewandowska D, Pazik J, Aveyard P, Stapleton J. Placebo-controlled trial of cytisine for smoking cessation. N Engl J Med. 2011 Sep 29;365(13):1193-200. doi: 10.1056/NEJMoa1102035. PMID 21991893
- [Background] Walker N, Howe C, Glover M, McRobbie H, Barnes J, Nosa V, Parag V, Bassett B, Bullen C. Cytisine versus nicotine for smoking cessation. N Engl J Med. 2014 Dec 18;371(25):2353-62. doi: 10.1056/NEJMoa1407764. PMID 25517706
- [Background] Walker N, Bullen C, Barnes J, McRobbie H, Tutka P, Raw M, Etter JF, Siddiqi K, Courtney RJ, Castaldelli-Maia JM, Selby P, Sheridan J, Rigotti NA. Getting cytisine licensed for use world-wide: a call to action. Addiction. 2016 Nov;111(11):1895-1898. doi: 10.1111/add.13464. Epub 2016 Jul 17. No abstract available. PMID 27426482
- See also: WHO report on the global tobacco epidemic, 2015 — http://apps.who.int/iris/bitstream/10665/178574/1/9789240694606_eng.pdf?ua=1&ua=1
- See also: Ministero della Salute, Istituto Superiore di Sanità. Linee guida cliniche per promuovere la cessazione dell'abitudine al fumo. Guida breve per la realizzazione degli interventi. — http://www.salute.gov.it/imgs/C_17_pubblicazioni_832_allegato.pdf
- See also: AIRC. Fumo: le domande più frequenti. Perché si insiste tanto sui rischi del fumo? — http://www.airc.it/prevenzione-tumore/fumo/tabagismo-smettere-fumare/